CLINICAL TRIAL: NCT02181933
Title: A Prospective Randomised Open Label Clinical Trial to Determine the Efficacy of Nevirapine, Compared With a Combination of ZDV + 3TC, in Decreasing the Peripartum Mother to Child Transmission of HIV. Women, Who Present After 38 Weeks Gestation or in Labour After 35 Weeks Gestation and Who Are Anti-retroviral Naive, Will be Included.
Brief Title: Efficacy of Nevirapine Compared to ZDV + 3TC Administered in Labor and Again at Postdelivery in HIV Positive Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1287
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine; Zidovudine; Lamivudine

ARMS (2):
- Nevirapine (Experimental): Mother: two doses, Infant: one dose
  Interventions: Drug: Nevirapine
- Zidovudine (ZDV) + Lamivudine (3TC) (Active Comparator)
  Interventions: Drug: Zidovudine (ZDV); Drug: Lamivudine (3TC)

INTERVENTIONS:
Drug: Nevirapine
  Arms: Nevirapine
Drug: Zidovudine (ZDV)
  Arms: Zidovudine (ZDV) + Lamivudine (3TC)
Drug: Lamivudine (3TC)
  Arms: Zidovudine (ZDV) + Lamivudine (3TC)

SUMMARY:
The primary objective of the study was to evaluate the efficacy of nevirapine versus ZDV+3TC (Zidovudine + Lamivudine), when administered in labor and again at postdelivery, in reducing peripartum mother to child transmission of HIV (Human Immunodeficiency Virus).

The secondary objective was to assess the overall HIV transmission rate between the 2 groups (intrauterine, intrapartum and postpartum up to 6 weeks) as well as to explore the relationship between infection and timing of maternal dose relative to birth, infant feeding method, maternal peripheral blood viral load, and other potential risk factors for transmission.

Following the introduction of the second and third Amendments to the Protocol, 2 substudies were added. The objectives of these substudies were to evaluate the frequency of resistance-conferring mutations to nevirapine (Amendment 2) and to ZDV+3TC (Amendment 3); to determine whether there was a reversion of any resistant virus to the wild type; and to determine if the resistant virus was transmitted from the mother to the child.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who present after 38 weeks gestation or in labour after 35 weeks gestation who are tested HIV positive. Estimated gestational age will be determined by one or more of the following:

  * Reliable menstrual history, which corresponds with uterine size
  * Physical examination
  * Estimated fetal weight
* A consent form for the mother and neonate will be signed by either the mother or the guardian prior to inclusion

Exclusion Criteria:

* Mothers who have taken any antiretrovirals in the last 12 months
* Mothers who are not able to take oral medication
* Mothers who present with ARDS (acute respiratory distress syndrome), septic shock or eclampsia
* Mothers presenting in discomfort, i.e. regular painful uterine contractions, or other factors that may contribute to her not being able to understand and sign the informed consent for HIV testing and study participation
* Use of another investigational drug or concurrent participation in another investigational protocol during the current pregnancy
* Unwillingness or inability to reasonably comply with the protocol (i.e., mother and neonate/infant could not be followed for the full 6 weeks of the trial)
* Grade 4 SGPT (Serum glutamate pyruvate transaminase) (>10 times the upper limit of normal value), if known prior to delivery
* A recent history (6 months preceding the study) or current evidence of drug abuse and/or alcoholism
* Mothers with fetuses with anomalies incompatible with life, if known prior to delivery
* Decision to deliver the infant by elective Cesarean section
* Amniocentesis was indicated
* Infants with severe growth retardation diagnosed before birth

Infants who fall into the following groups will not receive treatment, but the mother-infant pair will remain in the trial

* Infants with malformations incompatible with life
* Life-threatening perinatal conditions which do not allow oral therapy (e.g., sepsis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2648 (Actual)
Dates: Start 1999-04; Primary Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
Incidence of HIV transmission from a HIV positive mother to her exposed infant during the intrapartum and early postpartum period | Day 28, 42 and 56-84

SECONDARY OUTCOMES:
Overall HIV transmission rate (including intrauterine, intrapartum and postpartum) | up to 84 days
Time to infection | up to 84 days
Relationship between infection and timing of maternal dose relative to birth | up to 84 days
Relationship between infection and infant feeding method | up to 84 days
Relationship between infection and maternal peripheral blood viral load | Day 0 and 28
Relationship between infection and other potential risk factors | up to 84 days
Number of patients with adverse events | up to 84 days